CLINICAL TRIAL: NCT00497601
Title: A Prospective, Single Center, Open-Label, Dose-Escalation Phase II Study To Assess Safety and Efficacy Of Short-Course Regimens Of Amphotericin B Emulsion In Treatment Naïve Or Resistant Cases Of Visceral Leishmaniasis (Kala-Azar).
Brief Title: A Phase II Study To Assess Safety and Efficacy Of Short-Course Regimens Of Amphotericin B Emulsion In Kala-Azar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSV-AMBE II-KA-706
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral Leishmaniasis; Amphotericin B; Fat emulsion
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Amphotericin B; soybean oil, phospholipid emulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): Amphotericin B in fat emulsion (Amphomul) 7.5 mg/kg on day 1 and 3
  Interventions: Drug: Amphotericin B fat emulsion in visceral leishmaniasis; Drug: Amphotericin B fat emulsion; Drug: Amphotericin B in fat emulsion
- B (Experimental): Amphotericin B in fat emulsion (Amphomul) 10 mg/kg on day 1 and 5 mg/kg on day 3
  Interventions: Drug: Amphotericin B fat emulsion in visceral leishmaniasis; Drug: Amphotericin B fat emulsion; Drug: Amphotericin B in fat emulsion
- C (Experimental): Amphotericin B in fat emulsion (Amphomul) 12.5 mg/kg on day 1 and 2.5 mg/kg on day 3
  Interventions: Drug: Amphotericin B fat emulsion in visceral leishmaniasis; Drug: Amphotericin B fat emulsion; Drug: Amphotericin B in fat emulsion
- D (Experimental): Amphotericin B in fat emulsion (Amphomul) 15 mg/kg in a single dose administration on day 1
  Interventions: Drug: Amphotericin B fat emulsion in visceral leishmaniasis; Drug: Amphotericin B fat emulsion; Drug: Amphotericin B in fat emulsion

INTERVENTIONS:
Drug: Amphotericin B fat emulsion in visceral leishmaniasis — Amphotericin B in fat emulsion (Amphomul) 7.5 mg/kg on day 1 & 3 in group A Amphotericin B in fat emulsion (Amphomul) 10 & 5 mg/kg on day 1 & 3 in group B Amphotericin B in fat emulsion (Amphomul) 12.5 & 2.5 mg/kg on day 1 & 3 in group C Amphotericin B in fat emulsion (Amphomul) 15 mg/kg on day 1 in group D
  Other Names: Amphomul
Drug: Amphotericin B fat emulsion — Starting with 7.5 mg/kg on day 1 and 3, 10 and 5 mg/kg on day 1 and 3, 12.5 and 2.5 mg/kg on day 1 and 3 and finally 15 mg/kg on day 1
  Other Names: Amphomul
Drug: Amphotericin B in fat emulsion — Starting with 7.5 mg/kg on day 1 and 3, 10 and 5 mg/kg on day 1 and 3, 12.5 and 2.5 mg/kg on day 1 and 3 and finally 15 mg/kg on day 1
  Other Names: Amphomul

SUMMARY:
The purpose of this study is:

1. To evaluate the Safety and Efficacy of four different short-course regimens of Amphotericin B emulsion in treatment of Kala-azar (visceral leishmaniasis) subjects who are either treatment naive or treatment resistant to other antileishmanial drugs except amphotericin B containing preparations.
2. To assess the safety and efficacy of single-bolus infusion of Amphotericin B emulsion in treatment of Kala-azar.

DETAILED DESCRIPTION:
1. To evaluate the Safety and Efficacy of four different short-course regimens of Amphotericin B emulsion in treatment of Kala-azar (visceral leishmaniasis) subjects who are either treatment naive or treatment resistant to other antileishmanial drugs except amphotericin B containing preparations.
2. To assess the safety and efficacy of single-bolus infusion of Amphotericin B emulsion in treatment of Kala-azar.

Subjects will be administered the study drug in either of the following four dose levels in an ascending manner, starting with the first dosage regimen:

* 7.5 mg/kg on day 1 and day3 (Regimen 1)
* 10 mg/kg on day 1, followed by 5 mg/kg on day 3 (Regimen 2)
* 12.5 mg/kg on day 1, followed by 2.5 mg/kg on day 3 (Regimen 3)
* Single-bolus infusion of 15 mg/kg over 2-4 hours on day 1 (Regimen 4)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 years and 65 years of age (both inclusive).
2. Subject/subject's legally acceptable representative is willing and able to give written informed consent to participate in the study.
3. Treatment naive subjects having symptoms and/or signs of visceral leishmaniasis with parasitological confirmation of Kala-azar (by splenic or bone marrow aspirate smear examination).

If subjects are previously treated with other antileishmanial drugs except amphotericin B containing preparations, they will be enrolled in the study only after clinical and parasitological evidence that the disease is unresponsive to adequate treatment with other drugs, and after an appropriate wash out period

Exclusion Criteria:

1. Subjects with past history of treatment with Amphotericin B for Kala-azar.
2. Subjects positive for HIV infection.
3. Concomitant life threatening or serious disease.
4. Concurrent malaria (malarial parasite test to be negative prior to study treatment administration), tuberculosis or bacterial pneumonia.
5. Haemoglobin < 6 gm/dl, total leukocyte count < 1,500/cmm, platelet count < 50,000/cmm
6. Abnormal liver and renal functions (BUN and serum creatinine > 1.5 times upper limit of normal (ULN), AST/ALT > 2.5 times ULN, and bilirubin > 1.5 times ULN).
7. Pregnant or nursing women.
8. Known hypersensitivity to Amphotericin B or inactive ingredients of study drug formulation.
9. Subjects receiving any of the medications prohibited by the study protocol.
10. Evidence of significant haematological, cardiac, hepatic, renal, respiratory, neurological or metabolic disease or any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
11. Simultaneous participation in another trial or received any investigational product < 30 days prior to enrolment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Clinical and parasitological cure at end of treatment and final cure (no relapse) at six months, no hematological, hepatic or renal toxicity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, Principal Investigator — Banaras Hindu University
Locations (1):
- Kala-azar Medical Research Center, Muzaffarpur, Bihar, India